CLINICAL TRIAL: NCT02098954
Title: Second Line Erlitinib Combination With Gemcitabine Cisplatinum in Non-small Cell Lung Cancer Patients Who Harbored EGFR Sensitive Mutation Developed Resistance After First Line TKI Treatment
Brief Title: Erlotinib Combined With Chemotherapy in TKI Resistant Non-Small Cell Lung Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, HunanPTH, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKIRR001
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-Small Cell Lung; EGFR Gene Mutation
Keywords: TKI; resistance; erlotinib; combined chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): patients will received a 28 days gemcitabine platinum combined with erlotinib scheme(gemcitabine for day 1 and day 8, 1250mg/m2. Platinum for day 1, 75mg/m2. Erlotinib for 150mg/day, day 9-21 every cycle, after 4 cycles, erlotinib should be used daily), after 4 cycle of combined chemotherapy, patients will receive erlotinib for further treatment until progression disease.
  Interventions: Drug: Gemcitabine platinum combined with erlotinib

INTERVENTIONS:
Drug: Gemcitabine platinum combined with erlotinib — patients will received a 28 days gemcitabine platinum combined with erlotinib scheme, after 4 cycles combined chemotherapy, patients will receive erlotinib for maintain treatment until progression disease.Gemcitabine for day 1 and day 8, 1250mg/m2. Platinum for day 1, 75mg/m2. Erlotinib for day 9-21 during combined chemotherapy, 150mg/day, then erlotinib should be used daily until patients develop progression disease.
  Other Names: Gemzar; Tarceva

SUMMARY:
Numerous evidences verified that erlotinib could dramatically improve the PFS and OS of non-small cell lung cancers who harbor EGFR sensitive mutations, however, primary or secondary resistance will be developed after TKI treatment, doctors do plenty of researches to overcome TKI resistance. FAST ACT-2 study present that, first line erlotinib combined with chemotherapy could improved mOS to more than 30 months in NSCLCs who harbor EGFR sensitive mutations, several study shows that sensitive mutations still exist after TKI resistance, because of the next generation TKIs(such as BIBW2992) are not avaliable at present, agents for met amplification(such as Crizotinib) are so expensive that many Chinese patients could not support. Thus, the investigators hypothesis that, after first line TKI treatment, the patients who developed TKI resistance could still benefit from second line TKI combined with chemotherapy.

DETAILED DESCRIPTION:
The investigators will enroll patients diagnosed with advanced non-squamous,non-small cell lung cancer, patients with EGFR TKI sensitive mutations and developed TKI resistance in first line treatment. After enrollment, the investigators will do biopsy again before second line treatment to find out the potential mechanism of TKI resistance, do EGFR mutation test for both sensitive and resistant mutation in exon 18, 19, 20 and 21; do KRAS, BRAF and PI3K mutation test, do FISH for MET and HER-2, the investigators do all these test to evaluated both primary and secondary resistance, the investigators do all these tests to get an overview for EGFR mutation status of each patient who develop TKI resistance. For second line treatment, patients will received a 28 days gemcitabine platinum combined with erlotinib scheme, after 4 cycle of combined chemotherapy, patients will receive erlotinib for further treatment until progression disease. For the patients who have stable brain metastases, combined chemotherapy should begin after local treatment, such as whole brain radiotherapy or sterotactic radiosurgery.

the main endpoint of this study is mean PFS, second endpoints of this study consist of mean OS, 8 week ORR.

ELIGIBILITY:
Inclusion Criteria:

* advanced non-small cell lung cancer, stage IIIB/IV
* non-squamous
* EGFR sensitive mutations, such as exon 19 del, or exon 21 L858R
* received first line TKIs treatment and developed TKI resistance
* ECOG 0-2

Exclusion Criteria:

* squamous non-small cell lung cancer
* patients have unstable brain metastasis, predict survival less than 8 weeks
* spinal-cord compression without evidence of stabilisation or treatment
* women who were pregnant or lactating; women with a positive or no available pregnancy test result at baseline
* patients have any unstable illness that could not receive further treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
mean progression free survival(mPFS) | after patients receive treatment, mPFS should be measured before the third cycle of chemotherapy, after the fourth cycle, mPFS should be measured every 3 months up to two years
  mean progression free survival(mPFS) will be recorded in enroll patients who received second line gemcitabine platinum combined with erlotinib. mPFS should be measured before second line treatment, before the third combined chemotherapy, after the fourth combined chemotherapy, every 3 months during erlotinib treatment, mPFS should be measured up to two years or every time progression disease occurs within two years.

SECONDARY OUTCOMES:
mean overall survival(mOS) | every 3 months up to 3 years, or until all the survival data is obtained
  mOS should be measured since enrollment, every 3 months we will contact patients to find out detail survival data of each patient until 3 years, or within 3 years if all survival data is obtained.
8 week overall response rate(8 week ORR) | 8 week ORR should be measured after enrollment, the exact time point should be the ninth week after combined chemotherapy
  8 week ORR should be measured after enrollment, after combined chemotherapy for 8 weeks, the exact time point should be the ninth week during combined chemotherapy. CR, PR, SD shoud be measured according to RESICT 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Study Chair — Hunan Province Tumor Hospital
Locations (1):
- Hunan Province Tumor Hospital, Changsha, Hunan, China

REFERENCES:
- [Result] Wu YL, Lee JS, Thongprasert S, Yu CJ, Zhang L, Ladrera G, Srimuninnimit V, Sriuranpong V, Sandoval-Tan J, Zhu Y, Liao M, Zhou C, Pan H, Lee V, Chen YM, Sun Y, Margono B, Fuerte F, Chang GC, Seetalarom K, Wang J, Cheng A, Syahruddin E, Qian X, Ho J, Kurnianda J, Liu HE, Jin K, Truman M, Bara I, Mok T. Intercalated combination of chemotherapy and erlotinib for patients with advanced stage non-small-cell lung cancer (FASTACT-2): a randomised, double-blind trial. Lancet Oncol. 2013 Jul;14(8):777-86. doi: 10.1016/S1470-2045(13)70254-7. Epub 2013 Jun 17. PMID 23782814
- [Result] Suda K, Mizuuchi H, Maehara Y, Mitsudomi T. Acquired resistance mechanisms to tyrosine kinase inhibitors in lung cancer with activating epidermal growth factor receptor mutation--diversity, ductility, and destiny. Cancer Metastasis Rev. 2012 Dec;31(3-4):807-14. doi: 10.1007/s10555-012-9391-7. PMID 22736441